CLINICAL TRIAL: NCT00418275
Title: A Dose Finding, Pharmacokinetic and Safety Study of a Recombinant Human Plasminogen Activator (HTU-PA) in Patients With Acute Ischemic Stroke
Brief Title: Safety Study of a Recombinant Human Plasminogen Activator to Treat Acute Ischemic Stroke.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Global Biotech (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GB-001-P02
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2006-12

CONDITIONS: Cerebrovascular Accident
Keywords: Cerebrovascular Stroke
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Genetic: Recombinant Human Plasminogen Activator (HTUPA)

SUMMARY:
To evaluate the safety profiles of HTU-PA in patients with acute ischemic stroke.

DETAILED DESCRIPTION:
Cerebrovascular disease, the third leading cause of death after heart disease and cancer in developed countries, has an overall prevalence of 794 per 100,000. In the United States, it is estimated that more than 400,000 patients are discharged each year from hospitals after a stroke. The loss of these patients from the work force and the extended hospitalization they require during recovery make serious economic impact. In Taiwan, Cerebrovascular disease is the second cause of death.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with cerebral ischemia at any location producing a serious measurable deficit by NIHSS scale and who received study medication within 5 hours after the onset of the symptom. A serious measurable deficit by NIHSS was defined as the NIHSS  9 and  20 (for brain stem stroke, patients with NIHSS > 20 were included).
* Subjects were  18 years old, of either sex.
* Subjects or his/her legal guardians demonstrated their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Subjects with Modified Rankin Scale > 1.

Exclusion Criteria:

* Onset of symptoms on awaking from sleep.
* Intracranial bleeding detected on a pretreatment head computerized tomographic (CT) scan.
* Clinical presentation suggested a subarachnoid hemorrhage even if the head CT scan was normal.
* Head CT showed the evidence of early infarct sign > 1/3 of MCA territory.
* Subjects had generalized seizure at the onset of the stroke.
* Subjects with blood glucose < 50 mg/dl or > 400 mg/dl.
* Subjects had another stroke, head trauma, cerebral hemorrhage or ischemic infarction within 3 months prior to the study entry.
* Subjects with a significant surgery within 14 days prior to study entry.
* Subjects with a history of gastrointestinal or urinary tract hemorrhage within 21 days prior to the study entry.
* Subjects with lumbar puncture or arterial puncture of non-compressible site within 14 days prior to the study entry.
* Subjects had known bleeding diathesis.
* Subjects with other serious medical illness that interfered with the study.
* Subjects had a platelet count < 100,000/mm3; hematocrit < 30%.
* Subjects with other serious medical illness that interfered with the study.
* Subjects had aPTT or PT > upper normal limit.
* Subjects had uncontrolled hypertension (> 180 mmHg systolic or > 110 mmHg diastolic) without additional anti-hypertensive medication at screening visit.
* Subjects with recent transmural myocardial infarction and evidence of pericarditis within 3 weeks prior to the enrollment.
* Subjects had intracranial neoplasm, arteriovenous malformation, or aneurysm.
* Subjects had hemostasis defects including secondary to severe hepatic or renal disease.
* Subjects with history of drug or alcohol abuse within 1 year prior to the study entry.
* Subjects had significant hepatic dysfunction (SGOT/SGPT  3 x upper normal limit).
* Subjects had serum creatinine level  2 x upper normal limit or on renal dialysis.
* Subjects had administration of any other investigational drug within 30 days prior to study entry.
* Woman who was pregnant or nursing.
* Subjects had used other thrombolytics (streptokinase, tissue plasminogen activator, urokinase, anisoylated plasminogen streptokinase activator complex, anticoagulants).
* Subjects had severe cardiac disease (New York Heart Association Functional Classification III and IV).
* Subjects had history of cancer except inactive non-melanoma skin cancer, in situ carcinoma of the cervix, or any cancer in patient's disease free for more than 5 years.
* Subjects had any clinically significant deviation from normal in the physical examination that, in the investigator judgment, interfered with the study evaluation or affect subject safety.
* Subjects with history of lupus.
* Vasculitis was the cause of ischemic stroke.
* Subjects had been enrolled in this study previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2001-04; Study Completion 2004-06

PRIMARY OUTCOMES:
Major neurological improvement measured by NIHSS at 24 hours after treatment. "Major neurological improvement" is defined as 4-point improvement in the NIHSS measurement.

SECONDARY OUTCOMES:
Major neurological improvement measured by NIHSS at 30 minutes, 60 minutes, 2 hours, 48 hours, 7 days, 30 days, and 90 days after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Han-Hwa Hu, M.D., Study Chair — Taipei Veterans General Hospita-lNeurological Institute
Locations (1):
- Veterans General Hospita-lNeurological Institute, No. 201, Sec. 2, Shih-Pai Road, Taipei, Taiwan

REFERENCES:
- [Result] Hu HH, Teng MM, Hsu LC, Wong WJ, Wang LM, Luk YO, Chern CM, Soong BW, Sheng WY. A pilot study of a new thrombolytic agent for acute ischemic stroke in Taiwan within a five-hour window. Stroke. 2006 Mar;37(3):918-9. doi: 10.1161/01.STR.0000202591.18871.f7. Epub 2006 Jan 19. PMID 16424373